CLINICAL TRIAL: NCT06777576
Title: Empowering Mobility in People With Spinal Cord Injury With a Hands-free, Self-balancing Personal Exoskeleton
Brief Title: Self-balancing Personal Exoskeleton for SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wandercraft (Industry)
Collaborators: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP007
Record Dates: First submitted 2025-01-08; First posted 2025-01-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries (SCI); Paraplegia and Tetraplegia
Keywords: Spinal Cord Injury; Robotics; Community use; Hands-free exoskeleton; Overground exoskeleton; Walking; Self-balancing
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Hands-free exoskeleton (Experimental)
  Interventions: Device: Hands-free exoskeleton

INTERVENTIONS:
Device: Hands-free exoskeleton — A "device trainer specialist" from the investigation site will deliver training sessions with the exoskeleton to pair of participants (a pair corresponds to an individual with SCI and his/her companion). The device trainer will follow the progression of the pair through the training program and ensure they learn all the device "basic skills". Each training session lasts an average of 1.5 hours, variations according to the user's learning pace and tolerance. During the sessions with the exoskeleton, the participants will engage in mobility activities on different surfaces and perform Activities of Daily Living in simulated environments such as kitchen, bathroom, elevators and outdoor spaces.

SUMMARY:
This study aims to demonstrate the safety and effectiveness of the personal exoskeleton in individuals with spinal cord injury (SCI).

DETAILED DESCRIPTION:
This personal exoskeleton, developed by Wandercraft as a new version of the Atalante X, offers a novel hands-free and self-balancing design, aiming at enhancing stability and mobility for users in daily activities.

The study features an interventional, prospective, single-group, and open-label design, conducted over 3 to 4 weeks at two US research facilities. 24 subjects are required to complete the study. Anticipating a 15% dropout rate, the study will enroll 29 participants.

Over the course of nine to ten scheduled visits, participants undergo a sequence of procedures, beginning with screening and device fitting. This is followed by five training sessions which conclude with an evaluation to issue a competency certificate to confirm the ability to use the device across all its "basic skills". Additionally, two sessions are dedicated to evaluating the exoskeleton's effectiveness outcomes, complemented by an extra practice session. Each visit lasts an average of 1.5 hours.

ELIGIBILITY:
SCI user inclusion Criteria:

* Any gender, age 18 years or older;
* Motor complete or incomplete SCI with lesions at or above T6;
* ≥ 6 months post SCI;
* Able and willing to attend 9 to 10 visits1 to the center, including sessions of training and assessments of one-to-three hours duration;
* Able to read, understand, and provide informed consent;
* Living in the US and speaks English.

SCI user exclusion Criteria:

* Diagnosis of neurological injury other than SCI;
* Progressive condition that would be expected to result in changing neurological status;
* Severe concurrent medical disease, illness or condition judged to be contraindicated by the site physician;
* Unhealed or unstable traumatic or high impact lower extremity fracture of any duration that is, in the clinical judgement of the study physician, exclusionary for standing and walking;
* Knee (proximal tibia and/or distal femur) BMD <0.60 gm/cm2;
* Total hip BMD T-scores < -3.5;
* Fragility, minimal trauma, or low impact fracture of the lower extremity since SCI;
* Untreatable severe spasticity judged to be contraindicated by the site physician;
* Untreated/uncontrolled hypertension, as judged to be contraindicated by the site physician;
* Unresolved orthostatic hypotension (change from baseline seated BP to a fall in 20mmHg SBP and/or fall in 10mmHG DBP and symptoms when standing), or as judged to be contraindicated by the site physician;
* Open or unhealed skin pressure sores, abrasions, or bruises at any of the contact points of the exoskeleton;
* Morphological contraindications to the use of the device;
* Uncorrectable leg length discrepancy over 2 cm (about 0.79 in) when using additional correction tools;
* Unable to effectively operate the device with a hand-control interface, due to functional and/or cognitive impairment, evaluated based on the ability to manipulate the joystick in all direction, press and identify buttons on the hand control interface.
* Improper fitting in the device;
* Psychopathology documentation in the medical record that may conflict with study objectives;
* Pregnancy or women who plan to become pregnant during the study period;
* Concurrent participation in another interventional trial;
* History of uncontrolled autonomic dysreflexia;
* Presence colostomy and/or urostomy;
* Ventilator use at the time of the exoskeleton use.

Companion inclusion Criteria:

* Any gender, age 18 years or older;
* Willingness to attend 9 to 10 visits to the center, including sessions of training and assessments of one-to-three hours duration with the SCI user;
* Able to read, understand and provide informed consent;
* Living in the US and speaks English.

Companion exclusion Criteria:

* Inability to communicate with an assistant due to cognitive and language disorders;
* Any disease, concomitant injury, or condition that interferes with the performance or interpretation of the protocol- specified assessments;
* Insufficient strength and performance capability, evidenced by the ability to hold and retain the device in case of unbalance/fall;
* Insufficient availability to complete the study;
* Concurrent participation in another interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who complete the Timed Up and Go (TUG) in 3min or less. | At visit 7, after an average of 7.5 hours of training and at visit 9, after an average of 9 hours of training.
  The TUG evaluates the time from starting in a seated position to stand-up, walk 3 meters, turn around, walk back 3 meters and sit down on indoor surface.
Proportion of subjects who complete a distance of at least 40m on the Six-Minute Walk Test (6MWT). | At visit 7, after an average of 7.5 hours of training and at visit 9, after an average of 9 hours of training.
  The 6MWT measures the distance in meters traversed over 6 min, on indoor surface.

SECONDARY OUTCOMES:
Proportion of subjects who can complete at least 4 out of the 6 Activities of Daily Living (ADLs), in various simulated environments and with the exoskeleton. | At visit 7, after an average of 7.5 hours of training and at visit 9, after an average of 9 hours of training.
  The ADLs are done standing in front of the countertop in the kitchen, in a simulated living room, taking a 50m walk in the outdoor environment, taking the elevator, in the bathroom and walking in a hallway and through a door to get to the next room.
Proportion of subjects who complete the 10-Meter Walk Test (10MWT) on indoor surfaces in 1 minute or less. | At visit 7, after an average of 7.5 hours of training and at visit 9, after an average of 9 hours of training.
  The 10MWT measures the time in seconds taken to walk 10 meters.
Proportion of subjects who can don or doff the device within 10 minutes each, separately. | At visit 7, after an average of 7.5 hours of training and at visit 9, after an average of 9 hours of training.

OTHER OUTCOMES:
Proportion of users who pass the device "basic skills" certification evaluation at the end of visit 6. | Throughout the study and up until the end of Visit 6, after an average of 7.5 hours of training.
  During the Certification Evaluation, the users' performance in executing all the device usability critical tasks will be observed and assessed by the trainer to ensure they are performed correctly (i.e., executed safely, regardless of the level of companion assistance, that is documented but isn't a criterion for success). The "basic skills" certification evaluation is passed if all the device basic skills have been learnt through the previous training sessions with the device (visits 2-5) and the critical tasks are re-executed correctly during the evaluation at visit 6. The device basic skills cover device theoretical knowledge, proper setup and installation in the device, walking and other ambulatory functions on different surfaces, Activities of Daily Living in indoor and outdoor environment techniques on various surfaces, and safety features such as emergency extraction.
Number of users who successfully master the different basic skills at a given visit | Throughout the study and up until the end of Visit 6, after an average of 7.5 hours of training.
  For each basic skill, the visit number at which users are confirmed to have safely mastered the task is recorded on a "checklist", which lists all the device basic skills and is provided to the trainer. The goal is to track the users' learning progress and mastery of the device over time.
Evaluation of the assistance level provided by companion. | Throughout the study and up until the end of Visit 9, after an average of 9 hours of training and 3 hours of assessment.
  Assistance provided by the companion when mastering each basic skill on the checklist at initial learning, at the certification evaluation, during the additional practice session and when performing each test.
Overall Rating of Perceived Exertion (RPE) assessed with the Borg RPE scale by the users for the entire session. | At the end of visit 6 after an average of 7.5 hours of training, at the end of visit 7 after an average of 7.5 hours of training and 1.5 hours of assessment and at the end of visit 9, after an average of 9 hours of training and 3 hours of assessment.
  The Borg scale rates the perceived exertion between 6 and 20 (very very light to very very hard exertion). The SCI users and their companions are asked to give their rating for the entire session, separately.
Overall perceived safety with a 7-level Likert scale by the users on the entire session. | At the end of visit 6 after an average of 7.5 hours of training, at the end of visit 7 after an average of 7.5 hours of training and 1.5 hours of assessment and at the end of visit 9, after an average of 9 hours of training and 3 hours of assessment.
  Each participant - SCI user and companion separately - will be asked to provide his/her level of agreement on the following statement: "I felt safe during the session." by using a 7-level agreement scale from 1: "Strongly disagree" to 7: "Totally agree".
Up-right time in the device at each session | Throughout the study and up until the end of Visit 9, after an average of 9 hours of training and 3 hours of assessment.
  This measure is taken by the device itself.
Numbers of steps taken in the device at each session | Throughout the study and up until the end of Visit 9, after an average of 9 hours of training and 3 hours of assessment.
  The measure is taken by the device itself.
Distance walked in the device at each session | Throughout the study and up until the end of Visit 9, after an average of 9 hours of training and 3 hours of assessment.
  The measure is taken by the device itself.
Number of times the participants walk on each type of surface at each session | Throughout the study and up until the end of Visit 9, after an average of 9 hours of training and 3 hours of assessment.
  This data is collected by the device trainers at each session. Users are considered to have walked on a surface during a session if they have covered a minimum distance of 10 meters on that surface.
Perceived health benefits and overall satisfaction and motivation. | At visit 9, after an average of 9 hours of training and 3 hours of assessment.
  Perceived health benefits and overall satisfaction and motivation of the SCI users, assessed by a modified version of the Gagnon questionnaire.
  The statements under evaluation will be taken from the 41 statements originally found in the Gagnon questionnaire that encompass seven domains :
  * overall program satisfaction,
  * satisfaction with the robotic exoskeleton,
  * learnability of the robotic exoskeleton,
  * satisfaction with the program attributes,
  * perceived health benefits of walking with the robotic exoskeleton,
  * perceived risks and fears of walking with the robotic exoskeleton and
  * perceived motivation to engage in regular physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- James J. Peters, VA Medical Center, Bronx, NY, The Bronx, New York, United States